CLINICAL TRIAL: NCT05888051
Title: Age-related Differences on Low Back Pain and Lower Extremity Isokinetic Muscle Strength and Balance
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: E-10840098-772.02
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Back Pain
Keywords: balance
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young Adult
- Adult

SUMMARY:
Low back pain is one of the common problems that 80% of people experience at least once in their lifetime. Between 60% and 90% of the adult population are at risk for low back pain at some point in their lives. While most resolve within six weeks, relapses are common. Pain that lasts longer than 12 weeks is defined as chronic pain, and causes significant limitation in daily life and a high psychosocial burden due to pain. Chronic low back pain significantly limits occupational activities due to a decrease in functional status.

DETAILED DESCRIPTION:
Although chronic low back pain is a problem locally related to the lumbar and sacroiliac joints, it is also affected by changes in the joint and muscle structure of the lower extremity or affects these structures biomechanically. It has been shown that the endurance of the gluteus maximus muscle and the flexibility of the knee and hip flexors are decreased in individuals with chronic low back pain. Studies investigating knee extensor muscle strength in individuals with low back pain in the literature have shown that the maximum voluntary contraction of the knee extensors and the isokinetic strength of the knee extensors are decreased.

ELIGIBILITY:
Inclusion criteria;

* Being between the ages of 18 - 65,
* Volunteer. Exclusion criteria;
* Having a musculoskeletal or neuromuscular disease that limits mobility,
* Presence of lower extremity sequelae,
* Having undergone surgery on the Lumbar Region, having a history of systemic, inflammatory or cancer
* Participants of both genders will be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Participants; Questions will be asked in total, including information such as age, gender, height, weight, dominant hand.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | one day
  The most basic symptom seen in knee osteoarthritis is pain. As pain is a subjective sensation, it is often difficult to assess. Visual Analogue Scale, pain level, right and left extremities were evaluated separately. In addition, three different measurements were taken as rest, activity and night. For individuals, a value of 0 was "no pain"; A value of 10 was defined as "unbearably severe pain". The point marked by the patient was measured with a tape measure, and the examined value was recorded. Pain assessment was collected under three headings: at rest, during activity, and at night.
Lower Extremity Muscle Strength | one day
  In the measurement of lower extremity muscle strength, Quadriceps and Hamstring muscle strength will be measured with an isokinetic dynamometer (CSMI-Cybex Humac-Norm Testing & Rehabilitation System). The knee extension test will be performed in a sitting position. The test foot will be secured with a Velcro strap by placing it on the dynamometer arm 1 inch above the ankle. The lateral epicondyle of the femur will be used as the anatomical reference with which the axis of the dynamometer is aligned. Two different speeds of maximal reciprocal concentric isokinetic knee extension and flexion; It will be measured as slow (60°/s, 5 reps, 10 sec. rest) and fast (180°/s, 15 reps, 10 sec. rest).
Balance | one day
  Postural stability and joint movements decrease in patients with low back pain. The proper functioning of the musculoskeletal system is necessary to maintain postural control. In our study, we planned to evaluate the static and dynamic balance of the patients with the 'Biodex Balance System S.D.' balance and test device. This device; It is a device used to measure the stability limits of individuals, examining their balance abilities while trying to control and move the center of gravity on the support surface. This system has a mobile balance platform that can tilt its surface up to 20° in 360° range of motion. In this moving platform, 1 indicates the least stable level and 12 indicates the most stable level. This platform is linked to a computer software that allows the balance to be evaluated objectively.
Disability | one day
  The Oswestry Disability Index is a commonly used outcome measure to detect perceived disability in patients with low back pain. This index consists of 10 items, 8 of which are related to activities of daily living and 2 are related to pain. Each item is scored from 0 to 5, and the total score is expressed as a percentage, with higher scores corresponding to more disability). Increasing scores on the Oswestry Disability Index indicate a higher level of disability.

CONTACTS AND LOCATIONS:
Locations (1):
- HAZAL genç, Istanbul, None Selected, Turkey (Türkiye)

REFERENCES:
- [Background] Kim DH, Kim TH. Comparison of the effects of stability exercise and balance exercise on muscle activity in female patients with chronic low back pain. J Exerc Rehabil. 2018 Dec 27;14(6):1053-1058. doi: 10.12965/jer.1836438.219. eCollection 2018 Dec. PMID 30656169